CLINICAL TRIAL: NCT03597763
Title: Development of Persistent Fatigue Following Moderate and Severe Traumatic Brain Injury - Exploration of General and Injury-specific Mechanisms.
Brief Title: Fatigue Following Moderate and Severe TBI
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Extrastiftelsen (Other); Sunnaas Rehabilitation Hospital (Other); Personskadeforbundet LTN (Unknown); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Daniel Løke, Psychologist / PhD-candidate, University of Oslo
Other Study IDs: 2018/FO202360
Record Dates: First submitted 2018-07-02; First posted 2018-07-24 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Traumatic Brain Injury; Fatigue
Keywords: persistent fatigue; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological data will include standard blood test screening during hospitalization and 6 months follow-up, including tests to rule out other causes of fatigue: kidney, liver, thyroidal and pituitary status, haemoglobin, cortisol, B-12, D-vitamins and C-reactive protein (CRP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate to severe traumatic brain injury: Patients who have suffered a moderate to severe traumatic brain injury, with confirmed intracranial damage.

SUMMARY:
The subjective feeling of being periodically fatigued, tired, even exhausted is common in the general population, as well as in a large number of medical conditions, including neurological illness, such as traumatic brain injury (TBI), cerebrovascular accidents (CVA), multiple sclerosis (MS), and poliomyelitis. Fatigue typically results in compensatory behaviors such as spending extended time in bed, daytime napping, and restricted participation in activities of daily living, which in turn can have a profound negative impact on mental and physical health. Although fatigue is common and debilitating, there is a scarcity of knowledge concerning underlying biological, psychological and psychosocial mechanisms in the development and maintenance of persisting fatigue. There is also a general lack of theoretical accounts of potentially shared and etiology-specific mechanisms across conditions. The existence of clinical subgroups and diverse clinical trajectories is not well documented, resulting in a lack of evidence-based treatment opportunities. Diagnosis and management of fatigue is further challenged by difficulties in conceptualizing and defining the phenomenon itself, since fatigue is subjectively experienced and multifaceted. Thus, as fatigue often poses a chronic problem, health professionals in community based rehabilitation settings are faced with helping patients cope with this symptom without a clear understanding of causes or treatment options. The current project aims to map the occurrence of fatigue following moderate to severe TBI and achieve a better theoretical and clinical understanding of the mechanisms which may cause, exacerbate or protect against persisting fatigue following TBI. The study approach acknowledges that fatigue after neurological illness is the result of complex interplays between general individual predispositions and etiology-specific factors. A better understanding of these mechanisms is a prerequisite for personalized treatment and development of empirically based randomized controlled intervention studies. This approach has relevance to other clinical conditions as well. The long-term aim is to ensure accurate diagnosis, improve treatment and rehabilitation, and to contribute to knowledge based clinical decision-making both within specialized and community based rehabilitation settings.

DETAILED DESCRIPTION:
1.0. Fatigue following Traumatic Brain Injury (TBI) - definitions, measurement and prevalence.

Fatigue has been defined as "the awareness of a decreased capacity for physical and/or mental activity due to an imbalance in the availability, utilization and/or restoration of resources needed to perform an activity". TBI represents "an alteration in brain function, or other evidence of brain pathology, caused by an external force", and is among the most severe, disabling neurological disorders, with post-TBI fatigue (PTBIF) being one of the most common and debilitating chronic symptoms, regardless of injury severity. A challenge in studying PTBIF is related to difficulties in operationalization and assessment. Estimates of PTBIF rates thus vary from 21% to 73% due to heterogeneity of study populations, assessment strategies and study designs, e.g. time since injury, sampling of patients and fatigue measures employed. The numbers however typically by far exceed rates of fatigue in the general population, with one Norwegian study estimating 23%. Although numerous measures of fatigue exist, there is a lack of "gold standard" tools. Self-report instruments, VAS-scales and single item questionnaires are most common, and the Fatigue Severity Scale (FSS) has been documented to have good psychometric properties. There is however considerable overlap between measures of fatigue and other symptoms such as sleepiness, depression, and distress, resulting in less than optimal construct validity. Most studies of fatigue after TBI have furthermore used cross-sectional designs. Although very limited longitudinal data is available, there is some evidence to suggest that PTBIF levels may decline over the first 6 to 12 months post-injury, but remain steady or rise slightly thereafter. A recent study identified fatigue as the most common somatic complaint five years after TBI, affecting more than half of the patients. In summary, despite study variability, fatigue is a common and often chronic symptom after TBI. However, little longitudinal work has investigated individual variability in patterns of fatigue, rendering a lack of knowledge regarding sub-groups and clinical trajectories.

1.1. Contributing factors and theoretical accounts of PTBIF. Fatigue following TBI may be caused directly by the nervous system injury, i.e., primary fatigue, which is associated with deficits in cerebral networks mediating attention, arousal, and response speed (reticular activating system, limbic system, anterior cingulate, mid frontal, and basal ganglia). Primary fatigue may in turn be exacerbated by common symptoms after TBI, such as insomnia, pain, emotional distress, and reduced tolerance for physical and/or mental activity, i.e. secondary fatigue. Additional physical causes of PTBIF have also been noted, such as increased body mass index (BMI) leading to deconditioning, reduced physical activity and posttraumatic pituitary hormone deficiencies. Of notice, PTBIF does not seem to be related to the severity of injury as assessed by the Glasgow Coma Scale (GCS) or duration of post-traumatic amnesia (PTA). Ponsford et al. (2014) tested a model of the interrelationships between fatigue and daytime sleepiness, vigilance (i.e., sustained attention), anxiety, and depression after TBI. The findings indicated that fatigue after TBI is the precursor of anxiety, depression, and daytime sleepiness, and that fatigue exacerbates cognitive problems. However, this model needs to be replicated, as factors such as pre-and comorbid risk factors, premorbid fatigue, and personality were not included in the model, and the study used a cross-sectional design. The "coping hypothesis" put forward by van Zomeren and colleagues (1984) proposes that cognitive impairment, particularly reduced processing speed and attention, leads to a compensatory increase in brain activity and effort, which in turn results in fatigue. Some studies support this hypothesis, as increased brain (functional MRI) and autonomic reactivity (i.e., heart rate variability) was seen during cognitive effort in individuals with TBI compared to normal controls. Individuals with TBI have also been shown to experience greater fatigue while performing cognitive tasks requiring divided attention or other demanding cognitive processes. In their cost-benefit model, Boksem & Tops (2008) propose a theoretical framework emphasizing the role of automatic attributions of costs and benefits of mental and physical effort and rest in contributing to experienced fatigue. Mediated by dopaminergic structures, with medial frontal cortices playing a central role, it is proposed that heightened sensitivity to the short-term rewards of resting, in combination with a decreased sensitivity to the delayed rewards of long term goals, may lead to decreased intrinsic motivation to exert energy. Reward-related behavior is proposed to be associated with three factors; positive emotion towards the reward, a motivation to act in order to achieve it, and a capacity for learning stimulus-reward contingencies. An inverse relationship between self-reported reward sensitivity and fatigue has been reported in persons with Multiple Sclerosis, but no studies have explored the role of reward sensitivity PTBIF, despite the fact that both positive emotionality, motivated behavior and learning of reward contingencies are at risk of being affected by injury.

1.2. Risk factors for fatigue in the general population. In the general population, associations with fatigue have been found with demographic variables such as gender and educational level. Personality factors, such as neuroticism, have been linked to fatigue. Being high on neuroticism and perfectionism, and low on extraversion, constitute risk factors for experiencing exertion and fatigue, while extraverted people seem to be protected against high fatigue. Neuroticism might also moderate the role of catastrophizing cognitions and emotional distress on fatigue severity. Recent studies have also demonstrated that optimal levels of conscientiousness are related to a broad range of favorable health related behaviors and health outcomes, even including longevity. To our knowledge, conscientiousness, and personality in general, has not been much investigated in the context of PTBIF, nor in twin studies of fatigue. Emotional distress, anxiety and depression are commonly associated with fatigue, and may serve as both predisposing and perpetuating factors. Similarly, musculoskeletal pain, mood and sleep disturbances are associated with experienced fatigue in community dwelling adults.

In summary, there is reason to believe that individuals with TBI will be predisposed or vulnerable to develop PTBIF to variable degrees, as pre- and comorbid characteristics may act as both risk- and protective factors. Surprisingly, individual and general risk factors that may potentially contribute or even account for PTBIF, have not been extensively studied in populations with brain injury. Personality traits have been reported to be significant in mediating outcome following TBI, but the relationship between personality traits and persistent PTBIF has not previously been investigated.

2.0. Research Aims and Hypotheses. The primary aim of this study is to establish the frequency and severity of PTBIF in a representative sample of patients with moderate to severe TBI during the first year and a half post-injury, including investigation of potential clinical subgroups and trajectories of fatigue. We expect to find that fatigue will be a substantial and persisting problem for a large proportion of TBI patients. We furthermore hypothesize that there will be distinct clinical subgroups where the role of intra-individual factors such as premorbid fatigue, personality, somatic complaints, resilience, emotional distress, reward sensitivity and injury-related cognitive deficit will contribute differentially to persistent fatigue.

A secondary aim of the study is to explore the replicability of Ponsford´s (2014) model, wherein cognitive problems predicted fatigue, which in turn resulted in emotional distress. As we include a broader array of relevant individual factors, we hypothesize that the results will show multiple pathways to persistent fatigue, and expect to establish a more complex multidirectional model between the included factors.

3.0, Methodology. This longitudinal study takes on a broad clinical and theoretical perspective in exploring factors that might be predictive of persistent fatigue in a representative sample of patients with moderate-to-severe TBI over the first year and a half after injury, including comparison with a non-clinical twin-sample. A prospective longitudinal design will be applied, where a representative sample of patients with moderate and severe TBI will be assessed at 6 and 12 months post injury.

3.1. Statistical analyses and power. Analyses will be performed using the Statistical Package for the Social Sciences Version 22, with p<0.05 as level of significance. Change over time will be assessed using mixed models analysis at 3 time points: acute phase (T1), 6 months post-injury (T2), and 12 months post-injury (T3). Predictors of fatigue at 6 and 12 months post injury will be explored with linear regression analysis. The fatigue model presented by Ponsford et al. (2014) will be tested using path analysis, within a structural equation modelling framework. Based on previous reports, FSS scores ≥ 5 (on a scale ranging from 1-7) are interpreted as indicative of severe fatigue. According to the incident number of hospital-admitted adults with TBI in Eastern region of Norway, it is estimated that 130 patients with moderate-to-severe TBI, aged 18 - 65 years, will be eligible for study inclusion within one year. With an expected dropout rate of 20 - 30 %, we assume that 91-104 patients will be able to complete follow-ups. The statistical strength calculated with G*power 3.1.7 shows that a regression analysis with a correction for 10-13 predictors will yield a power of 81 % (effect size of 0.20, alpha of 0.05). One-point difference is a conservative indicator of an important change in individual FSS scores. Taking into account the total sample size, analysis of mean difference from T2 to T3 would permit a critical t of 1.98-1.99 and effect size of 0.28-0.30.

4.0. Plan for Activities, Visibility and Dissemination. Study results will be shared with the scientific community through scientific articles to be published in peer-reviewed international journals in the fields of neurology and rehabilitation, and through participation in scientific conferences. The PhD candidate will turn in his thesis containing three scientific articles addressing the study aims to the Department of psychology at the University of Oslo. Senior researchers in the group will publish additionally with him on the data set obtained in this study. Given the strong collaborative effort, the comprehensive data set, and the strong theoretical basis for this project, it has potential to result in high impact publications. Results will also be communicated through an ongoing dialogue with user organizations and central clinicians at Sunnaas Rehabilitation Hospital and Oslo University Hospital. A designated group of researchers and patient representatives within the project group will be responsible for planning of popularized presentation of results in order to communicate with society at large and to relevant patient groups. The research group will seek funding for hosting at least one large-scale scientific conference addressing mechanisms of fatigue in different clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe TBI (assessed by a Glasgow Coma Scale between 3-13 within the first 24 hours post-injury, and a radiologically confirmed intracranial injury)
* Patients from the Eastern part of Norway.

Exclusion Criteria:

* Pre- or comorbid neurological, medical or severe psychological disorders with the potential to cause fatigue.
* Ongoing substance abuse
* Cognitive or physical impairments to such a degree that neuropsychological assessment and self-report measures cannot be adequately applied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be identified through the collaboration with the Neurosurgical department at Ullevål, Oslo University Hospital (OUH), where the majority of patients in the Eastern part of Norway with moderate to severe traumatic brain injuries are admitted. Patients within our eligibility criteria are referred to Department of Physical Medicine and Rehabilitation at Ullevål, OUH. Some eligible patients not admitted to the Neurosurgical department, are routinely referred from other hospitals to Sunnaas Rehabilitation Hospital or Department of Physical Medicine and Rehabilitation at Ullevål, OUH. Patients are informed about the project by clinicians, and if they consent, the primary investigator contacts them to inform more thoroughly about the project. Patients who have been identified, but who do not arrive at clinical appointments, are sent an informational letter with an invitation to the project, with contact information.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 12 months post-injury
  A validated self-report questionnaire with norms available for the general Norwegian population, measuring primarily subjectively experienced functional consequences of fatigue. The scale provides a total average score of the nine Likert items ranging between 1-7, where 1 indicates little to no experienced functional limitations due to fatigue, and 7 indicates severe experienced functional limitations due to fatigue. The norms provide t-scores corrected for age, education and gender.
Chalder Fatigue Questionnaire | 12 months post-injury
  A validated self-report questionnaire with norms available for the general Norwegian population, with subscales for both mental and physical fatigue. The scale provides sum scores of mental (4 items), physical (7 items) and total fatigue, with individual items administered ranging between 0-3. High sum scores indicate higher degree of subjective fatigue. Norms provide t-scores corrected for gender and age on both subscales and the total score. In addition to the 11 items used to compute the subscale scores and the total score, two additional items address the longevity and extent of the subjective fatigue on a range between 0-3, where higher scores indicate longer duration of and more severe extent of the subjective fatigue problems.

SECONDARY OUTCOMES:
Giessen Symptoms Checklist - fatigue subscale | 12 months post-injury
  Subscale of the questionnaire measuring subjectively experienced fatigue, which provides an average score using six symptom items and reported symptom distress on a scale between 0-4 for both "in general" and "in the last two days".

OTHER OUTCOMES:
Giessen Symptoms Checklist | 6 and 12 months post-injury
  Self-reported subjective somatic symptom complaints. The questionnaire consists of 25 symptoms, and respondents are asked to rate the presence of each symptom on a scale of 0-4 "in general" and "in the last two days", thus providing a total of 50 responses. The responses provide average scores for the subscales of fatigue, gastrointestinal symptoms, musculoskeletal symptoms, cardio-vascular symptoms and a total average of subjective symptom distress.
Insomnia Severity Index | 6 and 12 months post-injury
  Self-reported sleep disturbances. The questionnaire consists of seven items rated on a scale of 0-4, where a higher sum score indicates more severe sleep disturbances.
Epworth Sleepiness Questionnaire | 6 and 12 months post-injury
  Self-reported sleepiness. The questionnaire consists of eight items rated on scale of 0-3, where a higher sum score indicates higher severity of problems relating to sleepiness.
The Behavioral Inhibition/Behavioral Activation Scale (BIS/BAS) | 6 and 12 months post-injury
  Self-report questionnaire assessing behavioral inhibition and activation traits. The questionnaire provides separate sum scales for Behavioral Activation (13 items) and its subscales Reward Responsiveness (5 items), Fun Seeking (4 items) and Drive (4 items), and a total sum score for Behavioral Inhibition (7 items). Each item is rated by the respondent on a scale between 1-4.
Pain drawing | 6 and 12 months post-injury
  Subjective reporting of pain-afflicted regions of the body, used to assess extent of pain.
Four NRS items on pain intensity | 6 and 12 months post-injury
  Four NRS items ranging 0-10 questioning namely the strongest and weakest pain intensity within the two last weeks, pain intensity in general, and pain intensity presently.
NEO Five Factor Inventory 3 | 6 and 12 months post-injury
  Personality assessment questionnaire, providing t-scores for the personality traits Openness, Conscientiousness, Agreeableness, Extroversion and Neuroticism. Respondents answer items ranging between 0-4, and sum scores are converted into scaled t-scores using the official norms corrected for gender.
Quality of Life after Brain Injury | 6 and 12 months post-injury
  Questionnaire specifically developed to measure fatigue in patients with acquired brain injury. The questionnaire provides scores for quality of life with regards to cognition (7 items), perception of self (7 items), daily life & autonomy (7 items), social relations (6 items), emotional status (5 items) and physical problems (5 items), as well as a total score (37 items). The average subscale and total scores are recalculated to a scale ranging between 0 and 100, where lesser scores indicate reduced quality of life.
Life Orientation Test Revised - Optimism subscale | 6 and 12 months post-injury
  Six selected items from the Optimism subscale to measure optimism as a trait, where individual items are rated on a scale of 0-4, and a higher average score indicates a higher degree of trait optimism.
University of California in Los Angeles (UCLA) Loneliness Scale | 6 and 12 months post-injury
  Three selected items from the questionnaire, where individual items are rated on a scale of 0-4, where a higher average scores indicate a higher degree of loneliness.
Rivermead Post-Concussion Questionnaire | 6 and 12 months post-injury
  Self-reported common somatic, emotional and cognitive symptoms following head injury, rated on a scale of 0-4, where 0 = no problems, 1 = symptom no longer a problem, and the ratings of 2-4 indicating higher degree of symptom burden. Sum scales are calculated for responses in the range 2-4 on the subscales of somatic (9 items), emotional (4 items) and cognitive (3 items) symptoms, as well as a scale for total symptom burden (16 items).
Resilience Scale for Adults | 6 and 12 months post-injury
  Self-report measure of various resilience factors. The questionnaire consists of 33 items rated on a scale between 1-5, with sum scores provided for the subscales Self Perception (6 items), Future Perception (4 items), Social Competence (6 items), Family Cohesion (6 items), Social Resources (7 items) and Structured Style (4 items), where higher sum scores indicate a higher degree of resilience.
Wechsler Abbreviated Scale of Intelligence (WASI) subtest - Similarities | 6 and 12 months post-injury
  Neuropsychological test of verbal abstraction abilities.
Wechsler Abbreviated Scale of Intelligence (WASI) subtest - Matrix Reasoning | 6 and 12 months post-injury
  Neuropsychological test of visual abstraction abilities and general intelligence.
Wechsler Abbreviated Scale of Intelligence (WASI) subtest - Vocabulary | 12 months post-injury
  Neuropsychological test of verbal comprehension and general intelligence.
Wechsler Adult Intelligence Scale IV (WAIS-IV) subtest - Digit span | 6 and 12 months post-injury
  Neuropsychological test of auditory attention and working memory.
Conners' Continuous Performance Test 3 | 6 and 12 months post-injury
  Neuropsychological test of sustained attention, vigilance and impulsivity
Delis-Kaplan Executive Function System (D-KEFS) subtest - Trail Making Test | 6 and 12 months post-injury
  Neuropsychological test of psychomotor speed and divided attention.
Delis-Kaplan Executive Function System (D-KEFS) subtest - Color Word Interference Test | 6 and 12 months post-injury
  Neuropsychological test of psychomotor speed, divided attention and impulse inhibition.
Iowa Gambling Task 2 | 12 months post-injury
  Neuropsychological test of decision making and reward/punishment sensitivity.
Cut Down, Annoyed, Guilty and Eye opener (CAGE) | 6 and 12 months post-injury
  Alcohol abuse screening tool consisting of four items where respondents are asked to indicate Yes or No to risk factors for alcohol abuse, with a sum score ranging between 0-4, where a higher score indicates higher risk of abuse. For this research project, additional questions are asked about whether these risk factors were also present premorbid to the injury.
Cut Down, Annoyed, Guilty and Eye opener, Adapted to Include Drugs (CAGE-AID) | 6 and 12 months post-injury
  Drug abuse screening tool consisting of four items where respondents are asked to indicate Yes or No to risk factors for drug abuse, with a sum score ranging between 0-4, where a higher score indicates higher risk of abuse. For this research project, additional questions are asked about whether these risk factors were also present premorbid to the injury.
Hopkins Symptoms Checklist 8 | 6 and 12 months post-injury
  Abbreviated research edition of the standardized inventory, used to assess depression and anxiety symptoms.
Negative Life Events Questionnaire | 6 and 12 months post-injury
  Self-reported negative life events last 12 months before injury, the first six months post-injury, and in the period between 6-12 months post-injury. Respondents are asked to indicate the presence or abscence of each of the 12 negative life events in these time periods, which provides a sum score of severe life events.
Two Numerical Rating Scale items about fatigue | 6 and 12 months post-injury
  One NRS item administered in advance of neuropsychological assessment (point 1), and one following assessment (point 2). The NRS items range between 1-10, where lower scores indicate a lower degree of experienced fatigue. Difference scores are computed by subtracting point 1 from point 2, and is used to measure perception of fatigability in the test situation.
Glasgow Outcome Scale Extended | 6 and 12 months post-injury
  Interview for categorizing functional outcome following traumatic brain injury. The interview provides a total score between 1-8, with the following categories: 1 = dead, 2 = Vegetative state, 3 = Severe disability, lower level, 4 = Severe disability, higher level, 5 = Moderate disability, lower level, 6 = Moderate disability, higher level, 7 = Good restitution, lower level, 8 = Good restitution, higher level.
Fatigue Severity Scale | 6 months post-injury
  A validated self-report questionnaire with norms available for the general Norwegian population, measuring primarily subjectively experienced functional consequences of fatigue. The scale provides a total average score of the nine Likert items ranging between 1-7, where 1 indicates little to no experienced functional limitations due to fatigue, and 7 indicates severe experienced functional limitations due to fatigue. The norms provide t-scores corrected for age, education and gender.
Chalder Fatigue Questionnaire | 6 months post-injury
  A validated self-report questionnaire with norms available for the general Norwegian population, with subscales for both mental and physical fatigue. The scale provides sum scores of mental (4 items), physical (7 items) and total fatigue, with individual items administered ranging between 0-3. High sum scores indicate higher degree of subjective fatigue. Norms provide t-scores corrected for gender and age on both subscales and the total score. In addition to the 11 items used to compute the subscale scores and the total score, two additional items address the longevity and extent of the subjective fatigue on a range between 0-3, where higher scores indicate longer duration of and more severe extent of the subjective fatigue problems.

CONTACTS AND LOCATIONS:
Overall Officials: Johan K. Stanghelle, Professor dr. med., Study Chair — Sunnaas Rehabilitation Hospital
Locations (2):
- Norway (2):
  - Sunnaas Rehabilitation Hospital, Nesoddtangen, Akershus
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Undecided